CLINICAL TRIAL: NCT00518843
Title: Family Therapy for Adolescent Bulimia Nervosa: A Controlled Comparison
Brief Title: Family Therapy for Adolescent Bulimia Nervosa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10208 (K23 MH01923)
Record Dates: First submitted 2007-08-17; First posted 2007-08-21 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Bulimia Nervosa
Keywords: binge eating; purging
MeSH Terms: conditions — Bulimia Nervosa; Bulimia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FBT-BN (Experimental): Family-based treatment
  Interventions: Behavioral: FBT-BN
- SPT (Active Comparator): Individual Supportive Psychotherapy
  Interventions: Behavioral: SPT

INTERVENTIONS:
Behavioral: FBT-BN — Mobilizing parents to curtail binge eating and purging
  Arms: FBT-BN
Behavioral: SPT — Supportive the individual patient to explore factors that might underlie the eating disorder
  Arms: SPT

SUMMARY:
The primary hypotheses are:

* A procedurally distinct family therapy is an effective and essential way to reduce bingeing and purging in adolescents with BN, and leads to the long-term amelioration of bulimic symptoms.
* Family therapy is an effective way to bring about meaningful improvements in family interaction.
* Family therapy will produce significantly larger reductions in bulimic symptoms and improved family interaction in adolescents with BN compared to a control supportive psychotherapy.

DETAILED DESCRIPTION:
Bulimia nervosa (BN) is a disabling eating disorder and affects as many as 2% of young women. It is a major source of psychiatric and medical morbidity that often impairs several areas of functioning. Even more alarming is the fact that BN is occurring with increasing frequency among adolescents and preadolescents. Applying stringent diagnostic criteria for BN, studies have found 2-5% of adolescent girls surveyed qualify for diagnosis of BN. Research specific to treatment of child and adolescent eating disorders remains limited. No psychological treatment has been systematically evaluated in the treatment of adolescents with BN. However, a series of studies from the Maudsley Hospital in London have shown that family therapy (the 'Maudsley Approach') is effective in the treatment of adolescents with anorexia nervosa (AN). These studies have shown that involving the parents and siblings in treatment has beneficial effects on reversing the course of the eating disorder as well as improving family interaction. A preliminary report from the Maudsley group has also shown that the 'Maudsley Approach' may be helpful in the treatment of adolescents with BN. Because most young adolescents still live with their families of origin, this raises the interesting clinical question that adolescent BN patients can also be successfully treated with family therapy.

The proposed study has two specific aims:

1. To adapt and pilot a recently developed family therapy manual for adolescent AN for use in the treatment of adolescent BN patients.
2. To compare the efficacy of this conceptually and procedurally distinct family therapy treatment with individual control psychotherapy.

To achieve these aims, we propose a five-year controlled treatment study to be carried out at The University of Chicago. Eighty newly referred adolescent patients meeting DSM-IV diagnostic criteria for BN will be randomly allocated to one of two groups: 1) family therapy or 2) the individual supportive control treatment. All patients will receive the same medical evaluation and monitoring throughout the study period. Assessment of psychiatric and medical outcome measures will be carried out at the onset of treatment, during treatment, at the end of treatment, and again at one-year follow-up. The clinical outcome variables assessed will include the EDE, KSADS, RSE, and EE.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV criteria for bulimia nervosa or partial bulimia nervosa

Exclusion Criteria:

* psychotic illness acute suicidality medical illness that impacts weight pregnant

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2001-04; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Binge eating and purging frequency measured by the Eating Disorder Examination | 28 days

SECONDARY OUTCOMES:
EDE Subscales | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Le Grange, PhD, Principal Investigator — The University of Chiacgo
Locations (1):
- The University of Chicago, Chicago, Illinois, United States